CLINICAL TRIAL: NCT00999596
Title: Clinical Image Evaluation Study for Philips MammoDiagnost DR Full Field Digital Mammography System (FFDM)
Brief Title: Image Evaluation of Philips Philips MammoDiagnost DR Full Field Digital Mammography System (FFDM)
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: PMSDR-2008-002 & 2010-002
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Digital Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- FFDM (Full Field Digital Mammography): Mammograms from the Philips Digital System

SUMMARY:
The purpose of this investigation, using hardcopy film, is to compare the accuracy of the Philips MammoDiagnost DR (FFDM device) and screen-film (SF) mammography in detection of breast cancer among women undergoing screening or diagnostic mammography.

Per the new FDA Guidance document for FFDM, accuracy in comparison to Screen-film is no longer required.

DETAILED DESCRIPTION:
The proposed research study is a prospective enriched reader trial in which patients who meet the study's eligibility criteria, subject to certain constraints specified in this protocol, will undergo both SF and the investigational Philips FFDM mammography. Two to five sites will participate as image acquisition centers. Images will be read by 9 mammographers reading the SF and Philips FFDM acquired images at various locations under the supervision of study managers.

Per the new FDA Guidance document for FFDM (Class II Special Controls Guidance Document: Full-Field Digital Mammography System), there is no longer a requirement for screen film images for a comparison and a reader study to determine accuracy is not required. 10 images acquired under protocols 2008-002a, 2010-002a and a European site will be read in a MQSA type study. This record has been modified to support the new FDA Guidance document.

The reviewers will evaluate the cases, using soft copy and hard copy images, noting the mammographic attributes for each case and documenting the findings on a clinical image evaluation form, which is very similar to what is used for MQSA Accreditation.

The following attributes will be assessed: in order to provide an overall assessment of whether these image sets collectively are of sufficient acceptable quality for mammography:

* Breast positioning, assessing coverage of the breast on craniocaudal(CC) and medio-lateral oblique (MLO) views, separately;
* Exposure, assessing visualization of the adipose and fibroglandular tissues and visualization of breast tissue underlying the pectoralis muscle, separately;
* Breast compression, assessing overlapping breast structures, uniformity of exposure of fibroglandular tissues, adequacy of penetration of thicker portions of the breast, exposure of thinner areas, and motion unsharpness;
* Image contrast for differentiation of subtle tissue density differences;
* Sharpness, assessing the edges of fine linear structures and tissues;
* Borders and benign calcifications;
* Tissue visibility at the skin line;
* Noise, i.e., noise obscuring breast structures or suggestive of structures not actually present;
* Artifacts due to image processing, detector failure and other factors external to the breast on hard-copy and soft-copy displays; and
* Overall clinical image quality

ELIGIBILITY:
Inclusion Criteria:

1. Patient underwent or is scheduled to undergo a screening or diagnostic mammogram examination (right and left craniocaudal and mediolateral oblique with or without special views) at one of the acquisition centers during the course of this research study.
2. At least 40 years of age
3. Provides written informed consent indicating willingness to participate in this research study prior to performance of the Philips FFDM mammogram
4. Meets none of the exclusion criteria

Exclusion Criteria:

1. Presence of a breast implant,
2. Patients undergoing a unilateral mammogram or an incomplete SF mammogram
3. had previously undergone an excisional breast biopsy
4. Pregnant women or patients who believe they may be pregnant

(f) Inmates (in accordance with 45 CFR 46.306)

(g) Patients who cannot, for any reason, undergo follow-up mammography examinations (where clinically indicated) at the participating institution

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening and diagnostic mammography patients
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Jalbert, Study Chair — Philips Healthcare
Locations (3):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
- Strahleninstitut CDT, Cologne, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated at out primary Diagnostic site in April 2010 and concluded in February 2011. A total of 35 diagnostic cases were obtained. Recruitment was initiated at out primary Screening site in May 2010 and concluded in November 2011. A total of 67 screening cases were obtained.
Pre-assignment Details: The trial was to evaluate performance of a FFDM system. During image acquisition FDA modified the trial criteria from an efficacy trial to a SE trial. Images from our diag site prior to Nov could not be used in this study as mag views were now required. Mag views were acquired in Jan-Feb 2011. Selected images were used from our screen site.
Period: Overall Study
Arm/Group | FFDM (Full Field Digital Mammography)
Started | 107
New FDA Guideline Released | 6 (FDA Guidance: Class II Special Controls Guidance Document: Full-Field Digital Mammography System)
Completed | 6 (Not all patient images were used for the reader evaluation based on new FDA Guidelines)
Not Completed | 101
Not completed — Statistical population not required | 101

BASELINE CHARACTERISTICS:
Arm/Group | FFDM (Full Field Digital Mammography)
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 104
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: FFDM (Full Field Digital Mammography) Mammogram Scores
Description: 6 mammography image sets (4 images per set) from women participating in the study were read and rated (pass/fail) by 2 MQSA (Mammorgraphy Quality Standards Act) certified mammography readers. A typical MQSA evaluation was performed on each image set and an image set was scored Pass or Fail. A total of 12 scores (6 image sets, 2 readers) were obtained.
Time Frame: Day 1
Population: This was not a statistical sample per FDA FFDM Guideline. FDA Guideline specified that a minimum of 6 film sets from the participants be analyzed. The number of participants required by FDA changed mid-study.
Measure: Number; unit: FFDM Mammogram set
Groups:
- FFDM Mammograms Score = Pass: Mammogram sets from the Philips Digital System with Pass score for Image Quality
- FFDM Mammograms Score = Fail: Mammogram sets from the Philips Digital System with Fail score for Image Quality
Arm/Group | FFDM Mammograms Score = Pass | FFDM Mammograms Score = Fail
Number analyzed (Participants) | 6 | 6
FFDM Mammogram set | 12 | 0

ADVERSE EVENTS:
Arm/Group | FFDM (Full Field Digital Mammography)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Change in requirements from FDA modified the reading study per the Nov 5, 2010 FDA Guideline for FFDM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less